CLINICAL TRIAL: NCT00296556
Title: A Randomized, Placebo-Controlled Trial of ONO-4819CD for Treatment of Mild to Moderate Ulcerative Colitis.
Brief Title: Therapeutic Study of ONO-4819CD for Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Collaborators: National Institute of Biomedical Innovation (Other Government)
Responsible Party: Hiroshi Nakase / Associate Professor, Kyoto University, Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRC05PG-II-1
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; EP4 agonist; PGE2
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rivenprost (drug)

SUMMARY:
The purpose of this study is to investigate whether ONO-4819CD is safe and effective in the treatment of mild to moderate ulcerative colitis.

DETAILED DESCRIPTION:
Ulcerative colitis is a relapsing disease of unknown cause characterized by bloody diarrhea. Therapy usually involves 5-aminosalicylates, corticosteroids and immunosuppressants. However, steroid resistance and dependency can become problematic. Immunosuppressive drugs, such as azathioprine, are beneficial but may have serious side effects. Therefore, new therapeutic approach is needed.

Prostaglandin E2 is one of the prostanoids, which is involved with innate immunity. PGE2 induces oral tolerance to specific antigen in the small intestine and downregulates the production and release of proinflammatory cytokines by macrophages and neutrophils. Accordingly, PGE2 is considered to be the mediator of mucosal protection.

Recently, it was elucidated that disruption of EP4 gene, which is one of PGE receptors, caused severe colitis in mice. Moreover, EP4-selective agonist (AE1-734) was also revealed to ameliorate severe dextran sodium sulfate-induced colitis in mice. We therefore examined the effects of 2 weeks intravenous EP4-selective agonist therapy for patients with mild to moderate ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ulcerative colitis
2. Mild to moderate ulcerative colitis refractory to 5-aminosalicylates therapy.
3. 20 years and above
4. Must obtain written informed consent

Exclusion Criteria:

1. Corticosteroids therapy within two weeks before enrollment
2. Immunosuppressive therapy within three months before enrollment
3. Leukocytapheresis therapy within one month before enrollment
4. Blood transfusion within two weeks before enrollment
5. Impaired renal function
6. Impaired hepatic function
7. Uncontrolled hypertension/hypotension
8. Uncontrolled arrhythmia
9. Impaired cardiac function
10. Cancer
11. Uncontrolled diabetes
12. Interstitial pneumonia
13. Glaucoma
14. History of colon resection
15. Infectious diseases needing medical treatments
16. Drug allergy
17. Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-02; Primary Completion 2007-12 (Estimated); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Remission evaluated by DAI scores at 14 and 28 days

SECONDARY OUTCOMES:
Improvement by DAI scores; Change in DAI scores; CAI scores at 3, 7, 14 and 28 days; Colonoscopic and histopathological scores at 14 and 28 days; Clinical severity and symptom scores at 7, 14 and 28 days; Cytokines at 7, 14 and 28 days; Adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Shuh Narumiya, MD, PhD, Study Chair — Kyoto University, Graduate School of Medicine; Tsutomu Chiba, MD, PhD, Principal Investigator — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University, Graduate School of Medicine, Kyoto, Japan

REFERENCES:
- [Background] Kabashima K, Saji T, Murata T, Nagamachi M, Matsuoka T, Segi E, Tsuboi K, Sugimoto Y, Kobayashi T, Miyachi Y, Ichikawa A, Narumiya S. The prostaglandin receptor EP4 suppresses colitis, mucosal damage and CD4 cell activation in the gut. J Clin Invest. 2002 Apr;109(7):883-93. doi: 10.1172/JCI14459. PMID 11927615
- [Background] Morimoto K, Sugimoto Y, Katsuyama M, Oida H, Tsuboi K, Kishi K, Kinoshita Y, Negishi M, Chiba T, Narumiya S, Ichikawa A. Cellular localization of mRNAs for prostaglandin E receptor subtypes in mouse gastrointestinal tract. Am J Physiol. 1997 Mar;272(3 Pt 1):G681-7. doi: 10.1152/ajpgi.1997.272.3.G681. PMID 9124591